CLINICAL TRIAL: NCT00846456
Title: Phase I/II Trial of Vaccine Therapy With Tumor Stem Cell Derived mRNA- Transfected Dendritic Cells in Patients Receiving Standard Therapy for Glioblastoma
Brief Title: Safe Study of Dendritic Cell (DC) Based Therapy Targeting Tumor Stem Cells in Glioblastoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Steinar Aamdal, Steinar Aamdal, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DC-CAST-GBM
Record Dates: First submitted 2009-02-15; First posted 2009-02-18 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Glioblastoma; Brain Tumor
Keywords: Tumor setm cell
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Dendritic cell vaccine with mRNA from tumor stem cells — Intradermal injection of transfected dendritic cells

SUMMARY:
The study induces an immune response towards the stem-cell like part of glioblastomas in combination with standard therapy. The aim is to define and characterize the feasibility, potential adverse effects of such therapy and measure time to progression and survival.

ELIGIBILITY:
Inclusion Criteria:

* Accessible volume and quality of tumor tissue for vaccine production
* MRI after surgery with minimal tumor remnant.
* Between 18 and 70 years of age.
* Must have histologically confirmed glioma grade IV, and a candidate for combined radiation therapy and chemotherapy ("Stupps regimen").
* Must be ambulatory with a ECOG performance status 0 or 1.
* A minimum 4 weeks must have elapsed between the end of glucocorticoid treatment and beginning of vaccination.
* Signed informed consent and expected cooperation of the patients for the treatment and follow up must be obtained and documented.

Exclusion Criteria:

* Tumor in a localization where a modest increase in size due to reactive oedema may have a large impact on patients neurological condition.
* Large tumor remnant after surgery.
* History of prior malignancy other than glioma, with the exception of curatively treated basal cell or squamous cell carcinoma of the skin and ca. cervicis stage IB.
* Chronic active infection requiring antibiotic therapy.
* Significant cardiac or other medical illness that would limit activity or survival, such as severe congestive heart failure, unstable angina, or serious cardiac arrhythmia.
* Prior splenectomy.
* Glucocorticoid treatment not possible to terminate due to autoimmune disease or increased intracranial pressure.
* Adverse reactions to vaccines such as asthma, anaphylaxis or other serious reactions.
* History of immunodeficiency or autoimmune disease such as rheumatoid arthritis, systemic lupus erythematosus, scleroderma, polymyositis- dermatomyositis, juvenile onset insulin dependent diabetes, or a vasculitic syndrome.
* Chemotherapy or other potentially immune-suppressive therapy that has been administered within 4 weeks prior to vaccination.
* Pregnancy or lactation.
* Any reason why, in the opinion of the investigator, the patient should not participate.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Adverse events | During follow-up

SECONDARY OUTCOMES:
Evaluation of immunological response, time to disease progression and survival time | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Steinar Aamdal, MD, PhD, Principal Investigator — Department of Clinical Cancer Research, Rikshospitalet; Iver A Langmoen, MD, PhD, Study Director — Dept of Neurosurgery, Ulleval University Hospital; Gunnar Kvalheim, MD, PhD, Study Director — Dept of cellular therapy, Rikshospitalet HF; Gustav Gaudernack, PhD, Study Director — Inst. of Immunotherapy, Rikshospitalet HF; Knut Lote, MD, PhD, Study Director — Dept. of oncology, Rikshospitalet HF; Jon Berg-Johnsen, MD, PhD, Study Director — Dept. of Neurosurgery, Rikshospitalet HF; Carl Langberg, MD, PhD, Study Director — Dept of oncology, Ulleval University Hospital; Marta Nyakas, MD, Study Director — Dept. of Clinical Cancer Research, Rikshospitalet HF; Einar O Vik-Mo, MD, Study Director — Dept of Neurosurgery, Ulleval University Hospital

REFERENCES:
- [Derived] Vik-Mo EO, Nyakas M, Mikkelsen BV, Moe MC, Due-Tonnesen P, Suso EM, Saeboe-Larssen S, Sandberg C, Brinchmann JE, Helseth E, Rasmussen AM, Lote K, Aamdal S, Gaudernack G, Kvalheim G, Langmoen IA. Therapeutic vaccination against autologous cancer stem cells with mRNA-transfected dendritic cells in patients with glioblastoma. Cancer Immunol Immunother. 2013 Sep;62(9):1499-509. doi: 10.1007/s00262-013-1453-3. Epub 2013 Jul 2. PMID 23817721